CLINICAL TRIAL: NCT03047187
Title: What is the Functional Status of Anterior Cruciate Ligament Reconstruction (ACLR) Patients at Discharge From Rehabilitation
Brief Title: The Functional Status of Anterior Cruciate Ligament Reconstruction (ACLR) Patients at Discharge From Rehabilitation
Acronym: SHOPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Husam Abdullah Almalki, Principal Investigator, University of Salford
Other Study IDs: 001
Record Dates: First submitted 2017-01-31; First posted 2017-02-08 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACLR patients: anterior cruciate ligament reconstruction patients
  Interventions: Diagnostic Test: ACLR

INTERVENTIONS:
Diagnostic Test: ACLR — * quadriceps and hamstring isometric muscles test
  * single hop for distance
  * IKDC, KOOS, Tampa and ACL-RSI Questionnaires

SUMMARY:
Objectives:

1. To examine the ability of ACLR patients at discharge from rehabilitation to perform a single-hop for distance.
2. To examine isometric muscle strength of ACLR patients at discharge from rehabilitation.
3. To examine ACLR patients' self-reported knee function at discharge from rehabilitation
4. To assess the psychological factors for ACLR patients at discharge from rehabilitation.
5. To correlate single-hop for distance with self-reported knee function, strength and psychological factors for ACLR patients at discharge from rehabilitation to discover whether any of these factors can predict the others.

DETAILED DESCRIPTION:
Aims:

1) To investigate subjective measures, objective measures, functional performance and psychological factors for ACLR patients at discharge from rehabilitation.

Hypothesis:

1-a There will be no differences between ACLR patients at discharge from rehabilitation, and return to sport criteria leg symmetry index (LSI ≥ 85%), in functional performance for single-hop for distance tests

1-b There will be no differences between ACLR patients at discharge from rehabilitation, and return to sport criteria leg symmetry index (LSI ≥ 85%), in objective measures of quadriceps and hamstring isometric muscle strength tests.

1-c There will be no differences between ACLR patients at discharge from rehabilitation, and return to sport criteria (LSI ≥ 85%) in subjective measures of self-reported knee function (KOOS) and (IKDC)

1-d There will be no differences in psychological factors for the anterior cruciate ligament return to sport after injury scale (ACL-RSI) between ACLR patients at discharge from rehabilitation and the cut-off score for return to sport (score ˃ 63).

1-e There will be no differences in the psychological factors for the Tampa scale of kinesiophobia between ACLR patients at discharge from rehabilitation and the cut-off score of fear of movement (score ≤ 37).

2) To investigate the relationship between self-reported knee function, isometric muscles strength, single-hop test and psychological factors post ACL reconstruction.

Hypothesis:

2-a There will be a correlation between self-reported knee function and isometric muscles strength in ACLR patients at discharge from rehabilitation.

2-b There will be a correlation between self-reported knee function and single-hop test in ACLR patients at discharge from rehabilitation.

2-c There will be a correlation between self-reported knee function and psychological factors in ACLR patients at discharge from rehabilitation.

2-d There will be a correlation between isometric muscles strength and single-hop test in ACLR patients at discharge from rehabilitation.

2-e There will be a correlation between isometric muscles strength and psychological factors in ACLR patients at discharge from rehabilitation.

2-f There will be a correlation between single-hop test and psychological factors in ACLR patients at discharge from rehabilitation.

Study Procedure After the participants confirm that they are interested in the study, they will be seen again at the rehabilitation class during their regular hospital appointment. During the participants' last visit to the rehabilitation department, they will be briefed again about the study, and if they agree to partake, they will be asked to sign the consent form.

Self-reported knee function The participants will be asked to complete the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire on symptoms, stiffness, pain, function daily living, function sport sand recreational activities and quality of life, and The International Knee Documentation Committee subjective knee form (IKDC) questionnaire, which assesses symptoms, function, and sports activity.

Psychological factors The participants will be asked to complete The Tampa Scale for Kinesiophobia (fear of movement) (TSK) which is a questionnaire that assesses pain related fear of movement followed by the Anterior Cruciate ligament Return to Sport after Injury (ACL-RSI) scales, which is a questionnaire that measures athletes' emotions, confidence in performance, and risk appraisal concerning to returning to sport following an ACL injury. A demographics form (age, height and weight) will also be completed.

Isometric muscle strength To gather isometric muscle strength data on each participant, data on isometric muscle strength for both legs will be obtained using two different tests for knee extensors and knee flexors muscles, using a hand-held dynamometer (HHD). The participants will be asked to wear sports clothing. The strength of both lower limbs of the participants will be assessed using the HHD, with peak force measured throughout five seconds of muscle contraction. Quadriceps muscles will be measured by first requesting the participants sit on the edge of the treatment bed with their knees 90 degrees flexion and both feet off the ground. The participants will then be asked to apply maximum force in extending the knee joint against the HHD device, which will be fixed using a belt and placed in front of the leg proximal to the ankle joint. They will be asked to do so for five seconds, and to repeat three times with 30 seconds of rest in between. The maximum peak force will be recorded throughout the three trials. To measure hamstring muscles, participants will be instructed to sit on the edge of the treatment bed with 90 degrees' flexion in the knee with both feet off the ground. Then, participants will be instructed to apply maximum force to flex knee joint against the immovable HHD device that will be fixed with a belt and placed at the back of the leg proximal to the ankle joint. They will be asked to so for five seconds, and this will be repeated three times with 30 seconds of rest in between. Maximum peak force will be recorded throughout the three trials.

Functional tasks Participants will be requested to perform a single-leg hop for distance, and this will be assessed using a standard metric tape measure. A 3m strip of tape will be placed on the floor, with the start line labelled using a 0.3m strip of tape placed perpendicular to the 3m strip of tape. The participants will be performed three practice trials for the hop test. After finishing the practice trials, four test trials will be asked to perform a single leg hop for distance as described by (Bolgla and Keskula, 1997). Attempts will be classified as successful provided the participant hops and lands with full stability on one leg for three seconds. The participants will be required to achieve four maximum hop attempts with complete stabilisation after landing for three seconds. Attempts will be deemed unsuccessful if the participant hops and touches the ground with their other leg during landing, or if they fail to hop within the limited marked distance; any failed hops will be counted and noted, but not processed. The participant's leg length will be measured while they are lying in a supine position before the first test using a standard tape measure to measure from the anterior superior iliac spine (ASIS) to the distal tip of the medial malleolus. Leg length will be used during data analysis to normalise excursion distances.

The participants will begin with their toe on the starting line, standing on one leg, before hopping as far as they can horizontally and landing on the same leg, and the distance hopped will be recorded. The hop data will be normalised to limb length by dividing the distance covered by the participant's leg length and then multiplying by 100, resulting in a percentage value. After completing the test, the participants will be asked to repeat the procedure with the other leg.

ELIGIBILITY:
Inclusion criteria:

In order to be eligible for the study they must meet the following:

1. Aged between 18 to 40 years old.
2. Adult with unilateral ACL injury and had an ACL reconstruction.
3. Subjects with no lower limb injury, pelvic or spinal pathology that limits the ability to hop comfortably.
4. They are confident they will be able to hop without an adverse reaction. This will be determined by the referring clinicians and approved the individual to hop.

Exclusion criteria:

Individuals who have any of the following will be excluded from the study:

1- Unable to give informed consent or comply with the study procedures. 2. Subjects with cardiovascular, pulmonary or neurological conditions that limited physical activity.

3. Subjects with any lower limb, pelvic or spinal pathology that limits the ability to hop comfortably.

4. Have not performed any hop landings during rehabilitation or have any apprehension about doing so

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited via orthopaedic consultants patient with unilateral ACL injury and had an ACL reconstruction. The principal investigator will organise to see the individual during their regular hospital appointment at the rehabilitation class to determine eligibility, then they will be briefed on the study and have all of the equipment and procedures explained to them. Any questions will be answered in full.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Hop test: by measuring the distance of single-hop for distance. | 12 months
  assessment of single hop for distance for ACLR patients at discharge from rehabilitation.

SECONDARY OUTCOMES:
Muscles strength: by measuring the peak force by using hand-held dynamometer | 12 months
  assessment of isometric quadriceps and hamstring muscles strength for ACLR patients at discharge from rehabilitation by using hand-held dynamometer.
Knee functions: by using (KOOS) | 12 months
  assessment of knee functions for ACLR patients at discharge from rehabilitation by using: The Knee injury and Osteoarthritis Outcome Score (KOOS).
Knee functions: by using (IKDC) | 12 months
  assessment of knee functions for ACLR patients at discharge from rehabilitation by using: The International Knee Documentation Committee (IKCD).
Fear of re-injury by using (TSK-17). | 12 months
  Assessment of fear of re-injury for ACLR patients at discharge from rehabilitation by using:
  TAMPA scale of kinesiophobia (TSK-17)
Readiness to return to sport after injury by using (ACL-RSI) scale. | 12 months
  Assessment of readiness to return to play after injury for ACLR patients at discharge from rehabilitation by using:
  Anterior Cruciate Ligament Return to Sports after Injury (ACL-RSI) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Herrington, PhD, Study Chair — University of Salford

IPD SHARING:
Plan to Share IPD: No